CLINICAL TRIAL: NCT06813469
Title: Multi-Dimensional Genomic Dissection of Ring Chromosome 14 Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MD-RING; RING 14 International Onlus (Other Grant/Funding Number: RING 14 International Onlus); PNRR-HEAL (Other Grant/Funding Number: MUR)
Record Dates: First submitted 2024-11-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Ring 14
Keywords: Ring14 Syndrome
MeSH Terms: conditions — Ring Chromosome 14 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lymphoblastoid Cell Lines (LCLs) (Other): 10 LCLs from r(14)S patients without other cytogenetic alterations were selected, as well as 5 LCLs from parents without cytogenetic alterations
  Interventions: Genetic: LRS analysis

INTERVENTIONS:
Genetic: LRS analysis — Long Read Sequencing (LRS) and High-throughput chromosome conformation capture (Hi-C) analysis to explore and functionally characterize the r(14) event and its impact on the three-dimensional (3D) genomic architecture inside the cells of r(14)S patients

SUMMARY:
MD-RING will explore the hypothesis that position effects and TAD alterations act as an unprecedented pathomechanism in r(14)S. This will contribute to a better understanding of genotype-to-phenotype correlations, creating an important scientific resource for the study of this and other ring syndromes, with the ultimate objective to offer improved family counseling , patient care and to identify potential new therapeutic options.

DETAILED DESCRIPTION:
Chromosome 14 ring syndrome [r(14)S] is a rare genetic disorder mainly characterized by complex and severe neurodevelopmental disorders, ranging from intellectual disability to aggressive/hyperactive behavior and drug-resistant epilepsy. Indeed, epilepsy is the most important clinical challenge in r(14)S, with enormous difficulty in controlling severe seizures and a strong need for innovative and effective treatments. Precision medicine for r(14)S patients would be greatly facilitated by knowledge of specific genes involved in pathogenesis. However, the pathophysiology of r(14)S is still largely unknown, and the identification of genotype/phenotype correlations is complicated by the co-occurrence of chromosome 14 rearrangements and the unknown degree of r(14) mosaicism in tissues most relevant to the disease. On the one hand, deletions of different sizes, from a few hundred Kbs to several Mbs, are often found in the terminal 14q region. These are an unlikely explanation for the severity and expressiveness of r(14) disease, since it has been observed that carriers of similar linear deletions of chromosome 14q rarely suffer from epilepsy. On the other hand, ring instability may promote increased monosomy of chromosome 14 in epilepsy-related areas of the brain (it is about 20% in peripheral blood).

Another fascinating hypothesis is that the mechanism and expressiveness of r(14) disease are driven primarily by the disruption of chromosome 14 conformation and positioning within the nucleus caused by its circularization, with dramatic effects on physiological interactions between genetic loci and, consequently, on gene regulation . This idea revives an unresolved question in cytogenetic disorders, whether the chromosomal abnormality itself produces a clinical phenotype beyond the pathogenic effects of the altered gene dosage. Rings can form from any chromosome, and most ring syndromes share largely similar clinical phenotypes. Severe epilepsy, for example, has been described in r(7), r(17), r(18), r(20), r(21) and r(22) syndromes in addition to r(14)S . This observation suggests that the presence of a loop within the nucleus may itself disrupt the balance of gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Ten LCLs of r(14)S patients with 14q deletions of varying position and extent in 70%, and monosomy 14 of varying degree in 60%.
* Five LCLs of parents without cytogenetic alterations.

Exclusion Criteria:

* Ten LCLs of r(14)S patients with 14q deletions of varying position and extent in 70%, and monosomy 14 of varying degree in 60%.
* Five LCLs of parents without cytogenetic alterations.

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
LRS analysis of SVs occurring on chromosome 14 | 8 months
  1. Resolving the sequence breakpoints of structural ring rearrangement in patients with r(14)S.
  2. Construct a 3D cell-specific molecular signature of r(14)S patients.
  3. Identify regulatory mechanisms that are important in the pathophysiology of r(14)S.

SECONDARY OUTCOMES:
Genotype-phenotype correlations based on the impact of the degree of mosaicism r(14) on the ability to identify Hi-C features. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Pippucci, Biologist, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No